CLINICAL TRIAL: NCT02376959
Title: Effect of Spiritist "Passe" Energy Therapy in Reducing Anxiety in Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associação Médico Espírita de Botucatu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31078414.5.0000.5411
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Complementary Therapies; energy therapies
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Application of 8 spiritist "passe" simulation sessions by people without spiritist training at the same time and in the same environment as the treatment group.
- Treatment Group (Spiritist "passe") (Active Comparator): Application of 8 sessions of spiritist "passe" by spiritists with more than 2 years of experience in controlled environments for the same period as the control group.
  Interventions: Behavioral: Spiritist "passe"

INTERVENTIONS:
Behavioral: Spiritist "passe" — For a period of 5 min per week, the volunteers will remain in the supine position with their eyes closed, in a quiet environment with controlled light and temperature.
  The applied intervention will consist of placing both hands in the classic Spiritist "passe" position for the stipulated 5-min period. Spiritist "passe" will be applied by volunteers with training and experience of more than two years with the technique.
  Arms: Treatment Group (Spiritist "passe")

SUMMARY:
Background: The use of alternative therapies in medicine has been increasing worldwide. Among these therapies are energy therapies such as Reiki , Johrei, and Spiritist "passe." Experimental studies have confirmed the action of the energy therapies in animal models or in cell cultures. These therapies appear to have positive effects, particularly in the reduction of anxiety and pain. Objective: To evaluate the effectiveness of the "passe" energy therapy in reducing anxiety in subjects presenting anxiety symptoms after 8 weeks of study. Methods: The recruited volunteers will be randomized into two groups: the Control Group (application of 8 "passe" simulation sessions by people without spiritualist training at the same time and in the same environment as the treatment group) and the Treatment Group (application of 8 sessions of "passe" by spiritists with over 2 years of experience in controlled environments for the same period as the control group). The sample will consist of 60 patients selected by interviews with the expectation of a 20% reduction of anxiety in the control group and 60% in the treatment group with alpha of 0.05 and beta of 0.8. Results: Using the STAI scale for evaluation, the reduction in anxiety is expected to be significantly higher in the treatment group than in the control group. The investigators expect approximately 20-30% reduction of the anxiety in the control group by the placebo effect. Other objectives to be assessed are quality of life, spirituality, and depression by specific standardized scales (WHOQOL-BREF, DUREL, and BECK).

DETAILED DESCRIPTION:
The use of complementary medicine has increased significantly worldwide and up to 40% of American patients use some form of complementary therapy[1,2 ]. Among these are the energy therapies such as Reiki[3], Johrei, and Spiritist "passe"[4]. These therapies are based on the modification of the energy fields that surround and penetrate the human body, and are supposedly involved in the health and disease process. Application of these therapies involves touch or laying hands on these energy fields, the existence of which has not yet been proven. Experimental studies have shown the action of energy therapies in animal models or in cell cultures[5,6,4]. Johrei proved to be effective in improving sleep in mice subjected to sleep interruption[5] and in reducing tumor cell growth in vitro[6]. An experimental study was recently published showing the effect of Spiritist "passe" on the growth of bacterial colonies of Escherichia coli. When "passe" was applied with the intention of reducing the growth of colonies there was a statistically significant reduction compared to the control group, subjected to laying of the hands without application of "passe" [4]. This study is recognized as the first experimental evidence of "passe" which is widespread in spiritism. Spiritism is a very common religion and philosophy in Brazil and the use of Spiritist "passe" is a form of treatment under this religion that is highly established in the treatment of psychiatric disorders[7,8]. Therapies used in spiritualism include Spiritist "passe," spiritist education, disobsession, and fluidic water. Studies investigating the scientific basis of these therapies are beginning to feature in the literature[8,9,10]. For energy therapies with clinical purposes, a few meta-analysis studies have evaluated distance healing and some touch therapies without reaching conclusive results, indicating a high heterogeneity between studies and presenting the need for more primary studies in the field[11,12]. Among the energy therapies, Reiki is the most widely studied; however, in recent meta-analysis, due to the large variability of the studies, different endpoints (anxiety, pain, depression) and methodological flaws, its efficacy has not yet been confirmed[13]. However, a more recent systematic review shows the efficacy of Reiki in reducing anxiety and pain[14].

Thus, despite the heterogeneity of the studies, energy therapies appear to have positive effects, particularly on the reduction of anxiety and pain. Spiritist "passe" is an important therapy in Brazil that is similar to other energy therapies such as Reiki and Johrei, and its efficacy has been experimentally confirmed[4]. Therefore, studies on clinical outcomes of this important form of complementary therapy are necessary. Unlike Reiki[14] and Johrei[15], there are no clinical studies on Spiritist "passe" despite its similar basis as an energy therapy.

1. STUDY HYPOTHESIS

The hypothesis of the study is that the Spiritist "passe" energy therapy will result in the reduction of anxiety, depressive symptoms, and improved quality of life in subjects with anxiety. The primary objective is to evaluate the Spiritist "passe" therapy in reducing anxiety in subjects with symptoms of anxiety after 8 weeks of study.

II. OBJECTIVES

1. PRIMARY OBJECTIVE

   The primary objective is to evaluate the efficacy of the Spiritist "passe" therapy in reducing anxiety after 8 weeks of study in subjects with symptoms of anxiety.
2. SECONDARY OBJECTIVES

   * Evaluate the impact of "passe" in reducing depressive symptoms
   * Evaluate the impact of "passe" on improving of quality of life
   * Evaluate the impact of "passe" on brain wave patterns detected with the electroencephalogram (EEG) III. PATIENTS AND METHODS

1. PATIENTS

1.1. Cohort:

Sixty patients with anxiety, who have not been treated by psychologists or doctors previously and do not use specific medication, will be evaluated. Patients will be recruited through the Botucatu Faculty of Medicine Press Service that will advertise phone numbers in newspapers and magazines and on the radio. Patients will be selected by the researchers according to the inclusion and exclusion criteria.

1.2. Outline: This is a randomized controlled prospective single-center study to evaluate the effect of Spiritist "passe" in reducing anxiety.

The trial will be conducted at a single location in the Clinical Hospital of the Botucatu Faculty of Medicine - UNESP.

Eligible patients who agree to participate and sign the informed consent form will be included in the study. The following four standardized questionnaires will then be administered:

1. DUREL questionnaire for assessment of spirituality
2. Beck Depression Inventory
3. State-Trait Anxiety Inventory (STAI)
4. WHOQOL-BREF quality of life questionnaire The questionnaires will be administered by an examiner who will read out the questions and write down the answers. The anxiety questionnaire (STAI) will always be administered first followed by the other questionnaires in random order.

After the questionnaires have been administered, patients will be randomly categorized into two groups, control and treatment (application of Spiritist "passe"), weekly according to the description of the study design.

1.3. Period: The study will begin after approval by the Research Ethics Committee of the Botucatu Faculty of Medicine. Thereafter, patients selected through interviews will be considered eligible if they meet the inclusion and exclusion criteria (described below in section 1.5). Eligible patients will be followed over an 8-week period with weekly applications of the treatment (Spiritist "passe") or the placebo (simulation of Spiritist "passe").

The standardized questionnaires will be administered three times (start, 4 weeks, and 8 weeks). Three assessments by electroencephalogram (start, 4 weeks, and 8 weeks) will also be made.

1.4. Sample: The sample will consist of 60 patients selected by interview following the inclusion and exclusion criteria. Based on the doctoral work of Ricardo Monezzi, the application of Reiki in elderly volunteers with stress resulted in a 20% reduction of anxiety level in the placebo group and 60% in the treatment group. Considering the reduction of anxiety in the control and treatment groups with an alpha of 0.05 and a beta of 0.8, respectively, a sample of 46 patients is planned. Assuming a 25% loss in follow-up, a sample of 60 patients is finalized.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater ≥18 years
2. Score of STAI-Trait questionnaire >41 (corresponding to the 51% for the Brazilian population)

Exclusion Criteria:

1. Patients with cognitive impairment who are unable to understand the questionnaires
2. Patients undergoing treatment for anxiety or depression
3. Patients undergoing psychological counseling
4. Patients receiving psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety questionnaire from baselaine at 8 weeks | Baselaine; 4 weeks and 8 weeks

SECONDARY OUTCOMES:
Change in Beck Depression Inventory from baselaine at 8 weeks | Baselaine; 4 weeks and 8 weeks
Change in WHOQOL-BREF quality of life questionnaire from baselaine at 8 weeks | Baselaine; 4 weeks and 8 weeks
Change in DUREL questionnaire for assessment of spirituality from baselaine at 8 weeks | Baselaine; 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Botucatu Medical School, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] de Souza Cavalcante R, Banin VB, de Moura Ribeiro Paula NA, Daher SR, Habermann MC, Habermann F, Bravin AM, da Silva CE, de Andrade LG. Effect of the Spiritist "passe" energy therapy in reducing anxiety in volunteers: A randomized controlled trial. Complement Ther Med. 2016 Aug;27:18-24. doi: 10.1016/j.ctim.2016.05.002. Epub 2016 May 6. PMID 27515871